CLINICAL TRIAL: NCT02387723
Title: Allogeneic Adipose Tissue-derived Stromal/Stem Cell Therapy in Patients With Ischemic Heart Disease and Heart Failure - a Safety Study
Brief Title: CSCC_ASC Therapy in Patients With Severe Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JKastrup (Other)
Responsible Party: Sponsor-Investigator, JKastrup, Professor Chief Physician, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCC_ASC1
Record Dates: First submitted 2014-12-29; First posted 2015-03-13 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem cell therapy (Experimental): Treatment with direct intra-myocardial Injection of 100 million allogeneic adipose derived stem cells (CSCC_ASC) into the heart
  Interventions: Biological: Allogeneic adipose derived stem cells (CSCC_ASC)

INTERVENTIONS:
Biological: Allogeneic adipose derived stem cells (CSCC_ASC) — Culture expanded allogeneic adipose derive stem cells (CSCC_ASC)

SUMMARY:
The present aim is to perform at small clinical safety trial in heart failure patients with allogeneic adipose tissue derived mesenchymal stem cells.

DETAILED DESCRIPTION:
Patients with heart failure will be treated with culture expanded adipose tissue derived mesenchymal stem cells from healthy donors stored in nitrogen until use. The cells will be injected directly into the myocardium using the NOGA XP method.

The patients will be followed for 6 months for safety and efficacy registration.

ELIGIBILITY:
Inclusion Criteria:

1. 30 to 80 years of age
2. Signed informed consent
3. Chronic stable IHD
4. HF (NYHA II-III)
5. LVEF ≤45%
6. Maximal tolerable angina and heart failure medication
7. Medication unchanged two months prior to inclusion
8. Angiography within six months of inclusion
9. No option for percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
10. Patients who have had PCI or CABG within six months of inclusion must have a new angiography less than one month before inclusion or at least four months after the intervention to rule out early restenosis
11. Patients cannot be included until six months after implantation of a cardiac resynchronisation therapy device

Exclusion Criteria:

1. Heart Failure (NYHA I or IV)
2. Acute coronary syndrome with elevation of CKMB or troponins, stroke or transitory cerebral ischemia within six weeks of inclusion
3. Other revascularisation treatment within four months of treatment
4. Moderate to severe valvular disease or valvular disease with option for valvular surgery
5. Diminished functional capacity for other reasons such as: coronary obstructive pulmonary disease (COPD) with forced expiratory volume (FEV) <1 L/min, moderate to severe claudication or morbid obesity
6. Clinical significant anaemia, leukopenia, leukocytosis or thrombocytopenia
7. Clinically significant abnormal prothrombin or partial thromboplastin time or anticoagulation treatment that cannot be paused during cell injections
8. Patients with reduced immune response or treated with immunosuppressive medication
9. History with malignant disease within five years of inclusion or suspected malignity - except treated skin cancer other than melanoma
10. Pregnant women
11. Other experimental treatment within four weeks of baseline tests
12. Participation in another intervention trial

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety: Number of patients with serious adverse events and development of tissue antibodies towards donor cells | 6 months
  Registration of number of patients with serious adverse events and development of tissue antibodies towards donor cells used for treatment in a 6 months follow-up period

SECONDARY OUTCOMES:
Cardial efficacy: left ventricle end-systolic volume (LVESV, ml), left ventricular ejection fraction (LVEF, %), end-diastolic volume (ml) and end-systolic mass (g) | 6 months
  The secondary objectives are to demonstrate improvement in in left ventricle end-systolic volume (LVESV, ml), left ventricular ejection fraction (LVEF, %), end-diastolic volume (ml) and end-systolic mass (g) between baseline and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, Professor MD, Study Director — Rigshospitalet, Denmark
Locations (1):
- 2014 Department of Cardiology, The Heart Centre, University Hospital Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared for Scientific collaboration